CLINICAL TRIAL: NCT06711497
Title: Global Postural Reeducation Exercises Versus Deep Neck Flexor Activation on Non Specific Neck Pain With Forward Head Posture
Acronym: GPR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: October 6 University (Other)
Responsible Party: Principal Investigator, Esraa Ahmed Mohamed Ahmed Mostafa, esraa ahmed mohamed ahmed, October 6 University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/005365
Record Dates: First submitted 2024-11-27; First posted 2024-12-02 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Non Specific Neck Pain; Forward Head Posture
Keywords: global postural reeducation; deep neck flexor activation; chronic non specific neck pain; forward head posture

STUDY DESIGN:
Intervention Model Description: global postural reeducation and deep neck flexor activation exercises
Who Masked: Participant, Outcomes Assessor
Masking Description: opaque sealed envelope
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- global postural reeducation exercise (Experimental): the patients will receive global postural reeducation and active neck flexor exercises twice a week for four weeks
  Interventions: Other: global postural reeducation exercises
- deep neck flexor activation exercise (Experimental): the patients will receive deep neck flexor activation with active neck exercises
  Interventions: Other: deep neck flexor activation exercise

INTERVENTIONS:
Other: global postural reeducation exercises — Subjects will be trained on global postural reeducation exercises (GPR) and active neck exercises. At each session, they will maintain two different lying postures to stretch anterior and posterior muscle chain and one standing posture to integrate the postural correction into activity of daily living (ADL.Initially, without gravity load, a lying posture was applied to the anterior muscle chain for approximately 15 min, then another lying posture to the posterior muscle chain for other 15 min, and finally the patients worked in a standing posture for postural integration under a gravity load for 5 min.
  Arms: global postural reeducation exercise
Other: deep neck flexor activation exercise — Subjects will be trained on deep neck flexor activation using pressure biofeedback and active neck exercises . The pressure sensor will be put under the neck and will be asked to de gentle nod as if saying "yes" so that the pressure sensor measures 2mmHg above baseline (20mmHg), then 4mmHg, followed by 6mmHg,8mmHg, and 10 mmHg without rests in between. the pressure sensor should read 30mmHg at the end of the movement sequence. Patient will hold each increment for 2 seconds, 10 seconds total after all 5 increments. Highest level achieved will be repeated with the correct form until a total of 10 reps with 10-second holds will be achieved in three series with 30 seconds of interval between the series plus active neck flexor exercise
  Arms: deep neck flexor activation exercise

SUMMARY:
this study will be conducted to compare between global postural reeducation (GPR) and deep neck flexors (DNF) activation in patients with chronic nonspecific neck pain (NSNP) on pain, disability, forward head posture and deep neck flexors endurance

DETAILED DESCRIPTION:
Neck pain (NP) is highly prevalent and is the sixth largest cause of disability in the world, causing considerable economic impact. Between 50% and 75% of people will not recover from an acute episode and will experience recurrent neck pain within the next 1 to 5 years, approximately 68% of people will develop persistent and chronic neck pain.Forward head posture (FHP) is a common posture malalignment which characterized by increased craniocervical angle more than 50 degrees. There is a significant association between neck pain and forward head posture. According to previous studies, it has been proven that an average of 60% of patients with neck pain have a forward head posture.Cranio-cervical flexor muscles training focuses on the deep flexor muscles such as longus capitis and longus colli muscles, which flex the neck, not the head. Also, these low-load exercises train the deep cervical flexors more specifically, rather than all the neck flexors involved in the head-lifting exercise.Global postural reeducation (GPR) is a method of physiotherapy, developed by Phillipe Souchard in the 1950s.Its therapeutic approach depends on causality, and globality and is based on the hypothesis that the muscular system is organized into muscle chains, which can be shortened because of musculoskeletal disorders and constitutional, behavioral and psychological factors. forty four patients will be assigned randomly into two equal groups; fist one will receive global postural reeducation plus active neck exercise and the other will receive deep neck flexor exercises plus active neck exercise

ELIGIBILITY:
Inclusion Criteria:

* Adult physiotherapists with mechanical neck pain and base line score of at least 3 out of 10 pain intensity on VAS .
* Adult physiotherapists with FHP and CVA less than 50 as a reference angle
* Adult physiotherapists aged from 18 to 24.

Exclusion Criteria:

* Specific cause of neck pain as (rheumatic ,sytemic ,neuromuscular diseases ).
* Cognitive impairment .
* Cervical radiculopathy .
* Cervical spondylolisthesis

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-02-15 (Estimated); Study Completion 2025-02-27 (Estimated)

PRIMARY OUTCOMES:
neck disability | up to four weeks
  neck disability will be measured by the Arabic version of neck disability index. NDI is a self-reported questionnaire that consists of 10 questions: pain intensity, personal care, lifting, reading, headaches, concentration, work, driving, sleeping, and recreation. Each item is scored from 0 (no disability) to 5 (total disability). The maximum possible score is 50. However, the NDI is frequently normalized to 100 and reported as percent Because the questionnaire is straightforward, most of the patients need approximately 5 minutes to complete it

SECONDARY OUTCOMES:
pain intensity | up to four weeks
  pain intensity will be measured by visual analogue scale. The VAS tool is a very simple tool as the therapist asks the patient to express how potent he/she feels current pain or last 24 hours' pain through choosing a point on a100 mm line drawn between two ends one end refer to absence of pain and the other the worst intense pain
Craniovertebral Angle | up to four weeks
  The Craniovertebral Angle will be measured using a digital imagining technique (kinovea software). The craniovertebral angle is measured by calculating the angle found at the intersection of a line drawn from the tragus of the ear through the spinous process of C7 Vertebra and a horizontal line through C7 Vertebra.
deep neck flexors endurance | up to four weeks
  deep neck flexor endurance will be measured by pressure biofeedback device. The pressure biofeedback unit will be centered just below the occiput between the plinth and the back of the neck and inflated to a baseline of 20 mmHg. Each subject was asked to execute the head nodding action gently and slowly (as if they said yes) at five different levels of pressure (22, 24, 26, 28 and 30 mmHg) and to maintain each level for 10 seconds There was a 30-second rest period between each level. The test protocol will end when the subject will be unable to hold the same pressure level for 10 sec or will reach a peak level of 30mmHg

IPD SHARING:
Plan to Share IPD: No